CLINICAL TRIAL: NCT04132609
Title: Opioid and Pain Cognitive Bias Modification in Opioid Use Disorder
Brief Title: Opioid and Pain Cognition
Acronym: opioid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2000024242
Record Dates: First submitted 2019-07-16; First posted 2019-10-21 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will complete the standard attentional bias task (control) or CBM up to 3x/week during MAT clinic visits for 4 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Intervention (Active Comparator): Complete cognitive bias intervention task during methadone clinic visit 3x/wk for 4 weeks.
  Interventions: Behavioral: Cognitive bias modification
- Control (Placebo Comparator): Complete standard attentional bias intervention task during methadone clinic visit 3x/wk for 4 weeks.
  Interventions: Behavioral: Standard attentional bias

INTERVENTIONS:
Behavioral: Cognitive bias modification — : In CBM, the task presentation and timing is the same as attentional bias, except the probe always replaces the neutral word. It ensures that: 1) the duration of CBM and control training should not differ; 2) CBM and control participants receive equal practice on the motoric aspects of the task; and 3) CBM and control participants are exposed to the same word cues. Based on previous data, duration of CBM and control trainings will be about 10 minutes.
  Other Names: Cognitive task
  Arms: Cognitive Bias Intervention
Behavioral: Standard attentional bias — the standard attentional bias task, a drug or pain-related word is presented next to a neutral word for 500ms. Subsequently, a probe (i.e., a "q" or "p") replaces the drug/pain word or the neutral word at an equal rate. The participant's task is to indicate the location of the probe as quickly as possible by pressing "q" or "p". Attentional bias is calculated from the difference in reaction times (i.e., neutral cue minus drug/pain cue) to indicate the location of the probe, with higher values indicating greater attentional bias. For all tasks, opioid and pain words will be presented in separate blocks in counterbalanced order. Neutral words paired with opioid or pain words will be matched for length and frequency of use in the English language.
  Other Names: Cognitive task
  Arms: Control

SUMMARY:
The proposed research will provide foundational research to develop this low-burden behavioral intervention that can potentially improve outcomes of OUD. The Specific Aims of the proposal include conducting a pilot randomized controlled trial with post-intervention and 3 month follow up to evaluate feasibility, acceptability, and preliminary effectiveness of CBM task for opioid and pain cues (Aim 1), examine naturalistic assessment of opioid craving and pain intensity/interference (Aim 2), and conduct qualitative analysis of Veterans experiences of adjunctive treatment in MAT clinic and perceptions of CBM as an intervention (Aim 3). Male and female Veterans meeting DSM5 criteria for OUD (N=60) currently on MAT will be randomly assigned to 4 weeks of CBM for opioid and pain cues or control (standard attentional bias). CBM/control tasks will be administered during weekly MAT clinic appointments and opioid craving and pain intensity/interference will be randomly assessed during the day using a mobile device. Post-intervention, Veterans will be invited to participate in a digitally recorded semi-structured interview for qualitative assessment of CBM and treatment adjunctive to MAT. MAT outcomes (urine toxicology screens, MAT appointments) will also be measured at 3-month follow up. The current study will elucidate dynamic relationships between attention to opioid and pain cues and whether modifying attention can reduce risk factors associated with treatment failure. If successful, with its low patient and provider burden, CBM could be readily incorporated in research and clinical practice as an adjunctive treatment for OUD.

DETAILED DESCRIPTION:
Participants will complete the standard attentional bias task (control) or CBM up to 3x/week during MAT clinic visits for 4 weeks.

Attentional bias: Attentional bias will be assessed during MAT clinic visits using the visual probe task, which is considered the gold standard to evaluate vigilance to salient cues. In the standard attentional bias task, a drug or pain-related word is presented next to a neutral word for 500ms. Subsequently, a probe (i.e., a "q" or "p") replaces the drug/pain word or the neutral word at an equal rate. The participant's task is to indicate the location of the probe as quickly as possible by pressing "q" or "p". Attentional bias is calculated from the difference in reaction times (i.e., neutral cue minus drug/pain cue) to indicate the location of the probe, with higher values indicating greater attentional bias. For all tasks, opioid and pain words will be presented in separate blocks in counterbalanced order. Neutral words paired with opioid or pain words will be matched for length and frequency of use in the English language. Opioid (e.g., syringe, needle, high, blues) and pain sensory (e.g., stuff, throbbing, shooting, burning) and affective (e.g., miserable, tiring, unbearable, exhausting) words will be taken from prior research demonstrating attentional bias in OUD and chronic pain patients.

CBM treatment: In CBM, the task presentation and timing is the same as attentional bias, except the probe always replaces the neutral word. It ensures that: 1) the duration of CBM and control training should not differ; 2) CBM and control participants receive equal practice on the motoric aspects of the task; and 3) CBM and control participants are exposed to the same word cues. Based on previous data, duration of CBM and control trainings will be about 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Veterans that meet DSM5 criteria for OUD
* Be engaged in Methadone Maintained Program
* Report clinically significant past-week pain intensity (i.e., at least moderate pain severity)

Exclusion Criteria:

* The inability to read, write and speak English
* Active suicidal ideation
* Diagnosis of psychotic disorder
* Use of drugs that interact negatively with MAT (e.g. benzodiazepines), and
* uncorrected defective vision, which would interfere completing the dot probe task

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Treatment-related Adverse events | 17 weeks
  The treatment-related adverse events will be measured as the number of participants assessed by cognitive behavior modification using an eprime task to compare the number of correct answers.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R MacLean, Ph.D., Principal Investigator — Yale University
Locations (1):
- Veteran Affairs Hospital, West Haven, Connecticut, United States